CLINICAL TRIAL: NCT05718492
Title: A Study of the Application of Hepatic Arterial Infusion in Advanced Hepatocellular Carcinoma Previously Treated With Immune Checkpoint Inhibitors and Antiangiogenic Agents
Brief Title: A Study of the Application of HAIC in Advanced HCC Previously Treated With ICIs and Antiangiogenic Agents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Zhao, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-508-01
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatic arterial infusion chemotherapy; Hepatocellular Carcinoma; Immunocheckpoint inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC (Experimental): Treated by HAIC alone.
  Interventions: Procedure: digital subtraction angiography.; Drug: FOLFOX (oxaliplatin , leucovorin , fluorouracil , and fluorouracil )

INTERVENTIONS:
Procedure: digital subtraction angiography. — Each patient received an artery catheter procedure guided by digital subtraction angiography.
Drug: FOLFOX (oxaliplatin , leucovorin , fluorouracil , and fluorouracil ) — Hepatic artery infusion chemotherapy. The FOLFOX (oxaliplatin 130 mg/m2, leucovorin 200 mg/m2, fluorouracil 400 mg/m2, and fluorouracil 2,400 mg/m2) regimen was sequentially infused through the catheter every cycle (3 weeks).

SUMMARY:
Immune checkpoint inhibitors (ICIs) plus antiangiogenic agents can achieve better efficacy than sorafenib in the treatment of hepatocellular carcinoma (HCC) within a certain period of time, but more than half of the patients are still insensitive to the treatment. There is no evidence-based basis for second-line treatment after the progression of the disease.In view of the effectiveness of Hepatic arterial infusion (HAIC) in the first-line treatment of HCC in the Chinese population, this study intends to launch a prospective intervention study to explore the efficacy and safety of HAIC treatment in patients with advanced HCC after the failure of ICIs and antiangiogenic agents combination therapy, and to provide high-level evidence for optimizing the second-line treatment of advanced HCC in the future.

DETAILED DESCRIPTION:
Each patient received an artery catheter procedure guided by digital subtraction angiography. Then, the FOLFOX (oxaliplatin 130 mg/m^2, leucovorin 200 mg/m^2, fluorouracil 400 mg/m^2, and fluorouracil 2,400 mg/m^2) regimen was sequentially infused through the catheter every cycle (3 weeks).A maximum of 4-6 courses of continuous hepatic artery infusion chemotherapy were received.If the patient has extrahepatic metastasis at baseline, ICIs should be used as a systemic treatment according to the severity of the disease. The drug type and treatment protocol of ICIs should be based on the most advanced treatment progress in the world.

ELIGIBILITY:
Inclusion Criteria:

Cytohistological confirmation is required for diagnosis of HCC. Patients with advanced (unresectable and/or metastatic, stage C based on Barcelona-Clinic Liver Cancer [BCLC] staging classification) hepatocellular carcinoma.

At least one tumor lesion meeting measurable disease criteria as determined by RECIST v1.1.

Current cirrhotic status of Child-Pugh class A-B, with no encephalopathy. Ascites controlled by diuretics is permitted in this study.

Availability of a representative tumor tissue specimen (archival tumor tissue is allowed) at pre-screening.

Eastern Cooperative Oncology Group Scale for Assessment of Patient Performance Status ≤ 2.

Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and 4 weeks after the completion of trial.

Adequate bone marrow, liver and renal function as assessed by central lab by means of the following laboratory requirements from samples within 7 days prior to procedure:

Hemoglobin > 100g/L Absolute neutrophil count >3.0 ×109/L Neutrophil count > 1.5 ×109/L Platelet count ≥ 50.0 ×109/L Total bilirubin < 51 μmol/L Alanine transaminase (ALT) and aminotransferase (AST) < 5 x upper limit of normal Albumin > 28 g/L Prothrombin time (PT)-international normalized ratio (INR) < 2.3, or PT < 6 seconds above control Serum creatinine < 110 μmol/L Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

Local treatments for HCC have been performed within 4 weeks, including surgical resection (including liver transplantation), local ablation, transcatheter arterial chemoembolization (TACE or TAE), radiotherapy (including brachytherapy).

A history of liver decompensation, such as refractory ascites, gastrointestinal bleeding, or hepatic encephalopathy; Uncontrolled complications, including but not limited to: Persistent or activity (except the HBV and HCV) infection, symptoms of congestive heart failure and uncontrolled diabetes, uncontrolled hypertension, unstable angina, uncontrolled arrhythmias, active ILD, severe chronic GI disease accompanied by diarrhea, or compliance with requirements may limit the research, resulted in significant increase risk of AE or influence Subjects provided psychiatric/social problem status on their ability to provide written informed consent. A history of active primary immunodeficiency or human immunodeficiency virus; Active or previous records of autoimmune disease or inflammatory diseases, including inflammatory bowel disease (e.g., colitis or Crohn's disease], diverticulitis, except [diverticulosis], systemic lupus erythematosus (SLE), sarcoidosis syndrome or Wegener syndrome (e.g., granulomatous vasculitis, gray's disease, rheumatoid arthritis, the pituitary gland inflammation and uveitis]).

Known to produce allergic or hypersensitive reactions to any study drug or any excipient thereof.

Significant clinical gastrointestinal bleeding or a potential risk of bleeding was identified by the investigator during the 30 days prior to study entry.

Tumors of the central nervous system, including metastatic brain tumors. Pregnant women or breast-feeding patients.

Complicated with other malignant tumors:

Malignant tumors that have been treated for therapeutic purposes, have no known active disease for 5 years prior to the first administration of the study drug, and have a low potential risk of recurrence.

Fully treated non-melanoma skin cancer or malignant freckle moles with no evidence of disease.

Fully treated carcinoma in situ without evidence of disease.

Is currently using, or has used an immunosuppressive drug within 14 days prior to the first dose of the investigational drug. This standard has the following exceptions:

intranasal, inhaled, topical or topical steroids. (e.g., intraarticular) Systemic corticosteroid therapy not exceeding 10 mg/ day of prednisone or its physiological equivalent as a prophylactic use of steroids for hypersensitivity. (e.g., CT scan pretherapy medication) Steroids as a prophylactic for allergic reactions. A live attenuated vaccine was administered within 30 days prior to the first administration of the study drug. Note: If enrolled, patients shall not receive live attenuated vaccine within 30 days of receiving study drug therapy and after the last administration of study drug.

Uncontrolled hypertension: systolic pressure ≥ 160 mmHg or diastolic pressure ≥ 100 mmHg despite anti-hypertension medications ≤ 28 days before randomization or first dose of drug.

Pregnant or lactating women, or fertile men or women who do not want to use high-efficiency contraceptives, 6 months after the last dosing of study treatment, from screening to study treatment. Based on the patient's preferred and customary lifestyle, abstinence during treatment and washout is an acceptable contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-10-18 (Estimated); Study Completion 2026-10-18 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2-years Followed up
  Tumor response to HAIC according to RECIST 1.1
Progress Free Survival (PFS) | 2-years Followed up
  Absence of disease progression other than death

SECONDARY OUTCOMES:
Overall Survival (OS) | 2-years Followed up
  Absence of death of any cause
Tumor local control | 2-years Followed up
  Absence of regrowth inside the treated lesion
Adverse Events (AEs) | 2-years Followed up
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhao, M.D. & Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Minimally Invasive and Interventional Radiology, Liver Cancer Study and Service Group, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lyu N, Wang X, Li JB, Lai JF, Chen QF, Li SL, Deng HJ, He M, Mu LW, Zhao M. Arterial Chemotherapy of Oxaliplatin Plus Fluorouracil Versus Sorafenib in Advanced Hepatocellular Carcinoma: A Biomolecular Exploratory, Randomized, Phase III Trial (FOHAIC-1). J Clin Oncol. 2022 Feb 10;40(5):468-480. doi: 10.1200/JCO.21.01963. Epub 2021 Dec 14. PMID 34905388
- [Result] Lyu N, Kong Y, Mu L, Lin Y, Li J, Liu Y, Zhang Z, Zheng L, Deng H, Li S, Xie Q, Guo R, Shi M, Xu L, Cai X, Wu P, Zhao M. Hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin vs. sorafenib for advanced hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):60-69. doi: 10.1016/j.jhep.2018.02.008. Epub 2018 Feb 20. PMID 29471013
- [Result] Lyu N, Lin Y, Kong Y, Zhang Z, Liu L, Zheng L, Mu L, Wang J, Li X, Pan T, Xie Q, Liu Y, Lin A, Wu P, Zhao M. FOXAI: a phase II trial evaluating the efficacy and safety of hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin for advanced hepatocellular carcinoma. Gut. 2018 Feb;67(2):395-396. doi: 10.1136/gutjnl-2017-314138. Epub 2017 Jun 7. No abstract available. PMID 28592441